CLINICAL TRIAL: NCT05951504
Title: The Prospective Evaluation of Peri-Operative Glucocorticoid Use in the Management of Cervicofacial Infections of Odontogenic Origin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ryan McCoy, DDS, Oral and Maxillofacial Surgery Resident, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS25101
Record Dates: First submitted 2023-07-04; First posted 2023-07-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Odontogenic Infection of Jaw (Disorder)
Keywords: Glucocorticoid
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Solumedrol 1 Dose (Active Comparator): Patients with an odontogenic cervicofacial infection were treated with one dose of Solumedrol 125mg intravenous at time of surgery. Remainder of management was as per protocol.
  Interventions: Drug: Methylprednisolone
- Solumedrol 4 Dose (Active Comparator): Patients with an odontogenic cervicofacial infection were treated with one dose of Solumedrol 125mg intravenous at time of surgery, as well as three consecutive doses of Solumedrol 125mg intravenous every six hours post-operatively. Remainder of management was as per protocol.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Patients with an odontogenic cervicofacial infection were randomized between two intervention groups. Patients in one group were treated with one dose of Solumedrol 125mg intravenous at time of surgery. Patients with an odontogenic cervicofacial infection in the other group were treated with one dose of Solumedrol 125mg intravenous at time of surgery, as well as three consecutive doses of Solumedrol 125mg intravenous every six hours post-operatively. Remainder of management was as per protocol.
  Other Names: Solumedrol

SUMMARY:
This study is a clinical trial. In Manitoba, the treatment of cervicofacial infections of odontogenic origin which require inpatient medical and surgical management by Oral and Maxillofacial Surgeons are treated in a reproducible and stepwise manner. After a standardized pre-operative diagnostic workup (including appropriate imaging, bloodwork, and pre-operative history and physical), these patients are taken to the operating room for appropriate surgical intervention (extraction of necessary teeth and incision/drainage of the associated abscess). These patients are then treated with a combination of antibiotics, steroids, and adjunctive medications as needed for supportive care until ready for discharge.

Intravenous corticosteroids are frequently administered following dentoalveolar and maxillofacial surgery procedures to decrease post-operative edema, improve patient comfort, and thus hasten recovery time. Within the context of primary and deep space odontogenic infections, one of the major sources of morbidity is the mass effect produced by edema causing airway obstruction. Additionally, manipulation of the soft tissues during the surgical procedure(s) (incision and drainage, extraction of teeth, etc.) may result in increased swelling around the airway. Inflammation and spasm of the muscles of mastication is another sequelae of infection, which can result in severe trismus. The literature supports the use of intravenous corticosteroids as an adjunctive treatment in the management of primary and deep space neck infections, and thus corticosteroid use is within the standard of care. However, the glucocorticoid dosing regimen is currently determined by the clinical judgment of the attending surgeon. One commonly used regimen for steroid dosing is prescribing Solumedrol 125mg IV X1 dose at the time of surgery. Another commonly used regimen for steroid dosing is prescribing Solumedrol 125mg IV X1 dose at the time of surgery, followed by 3 consecutive doses of Solumedrol 125mg IV every 6 hours post-operatively.

The goal of this study is to guide future decisions related to the treatment of patients with cervicofacial infections of odontogenic origin in Manitoba. This study is intended to follow the post-operative inpatient course of 30 patients with various cervicofacial infections of odontogenic origin. All will be treated via a standardized surgical protocol (incision/drainage and extraction of necessary teeth), antibiotics, and steroids. 15 patients will be randomly assigned to receive 1 dose of Solumedrol 125mg IV at the time of surgery but no doses following surgery. The remaining 15 patients will receive 1 dose of Solumedrol 125mg IV at the time of surgery plus 3 consecutive doses of Solumedrol 125mg IV every 6 hours post-operatively. In summary, the only impact of study involvement will be the determination of the intravenous glucocorticoid dosing schedule, as all patients will continue to receive the current standard of care (including surgical management, antibiotics, and intravenous corticosteroids).

To ensure the preservation of the highest level of patient care, in the rare instance where an attending surgeon decides peri-operatively that the pre-determined steroid dosing regimen will result in unsatisfactory treatment, the randomized patient assignment will be abandoned, and alternative treatment regimens will be used under the guidance of the attending Oral and Maxillofacial Surgeon.

Treatment will be undertaken at the Health Sciences Centre adult operating room and inpatient wards, the primary operating site for the University of Manitoba's attending on-call Oral and Maxillofacial Surgeons. The patient's post-operative course in hospital will be completed within the inpatient wards at the Health Sciences Centre, until the patients are deemed appropriate for discharge.

Specific patient outcomes will be evaluated at the time of hospital admission, daily while admitted to hospital, and at the time of hospital discharge. Outcomes evaluated will include:

* C reactive protein (CRP) levels (acute phase reactant which is a hematologic biomarker of inflammation)
* White blood cell (WBC) levels (hematologic biomarker of infection)
* Length of hospital admission (days)
* Trismus (in mm)
* Daily clinical examination findings (during morning inpatient rounds while admitted)

This study poses no additional risks to the patients involved, as these patients would be receiving intravenous glucocorticoids whether they were enrolled in the study or not. There are standard risks of complications involved with both the surgical and pharmaceutical treatment of cervicofacial infections of odontogenic origin, and these risks are discussed with patients pre-operatively and prior to hospital admission to obtain informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over the age of 18 years old
* Patients with a cervicofacial infection of odontogenic origin that require hospital admission and surgical intervention under the care of the Oral and Maxillofacial Surgery Department at Health Sciences Centre, and a post-operative course in hospital until such time that the patient is deemed suitable for discharge

Exclusion Criteria:

* Patients in whom consent for treatment of cervicofacial infections of odontogenic origin is not obtained pre-operatively, either by the patient or an appropriate alternative decision maker. Patients at the Health Sciences Centre are required to sign their own consent, or in the case of patients unable to sign their own consent for legal or medical reasons, an alternative decision maker is required to provide consent prior to undergoing treatment under general anesthesia/admission (this includes the administration of steroids at the time of surgical intervention and post-operatively)
* Patients with pertinent medical history that precludes the use of high-dose steroids, including: known hypersensitivity to steroids, severe immune compromise precluding the use of steroids, poorly controlled Type 1 diabetic patients, systemic fungal infections, latent tuberculosis, herpes simplex keratitis, acute psychosis, Cushing's syndrome, peptic ulcer disease, pregnant patients, breastfeeding mothers, markedly elevated creatinine/significant renal disease
* Patients with concomitant facial fractures leading to cervicofacial infections
* Patients with pathologic soft tissue or bony entities leading to cervicofacial infections
* Patients with cervicofacial infections of non-odontogenic origin (where adequate source control may be unachievable)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Admission | Entire length of hospital admission (in days), total average length less than 14 days
  Length of Hospital Admission in days from the date of admission to the date of discharge.
White Blood Cell Count | Daily for entire length of hospital admission (in days), total average length less than 14 days
  Hematologic Biomarker of Infection
C-Reactive Protein Level | Daily for entire length of hospital admission (in days), total average length less than 14 days
  Acute phase reactant that is a hematologic biomarker of infection
Improvement in Mouth Opening (Trismus) | Daily for entire length of hospital admission (in days), total average length less than 14 days
  Trismus is a marker of both pain and resolution of soft tissue swelling

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCoy, DDS, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No